CLINICAL TRIAL: NCT03805568
Title: The Effect of Dexmedetomidine and Remifentanil on the Postoperative Sore Throat After Thyroidectomy
Brief Title: A Postoperative Sore Throat After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-03-037
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Post Operative Sore Throat
Keywords: postoperative sore throat; dexmedetomidine; remifentanil; thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine infusion group (Active Comparator): dexmedetomidine infusion (loading dose of 1 ㎍/kg over 10 min and continuous infusion of 0.3-0.6 ㎍/kg/h) during the surgery
  Interventions: Drug: dexmedetomidine infusion group
- remifentanil infusion group (Active Comparator): remifentanil of 4 ng/ml during induction, followed by remifentanil infusion (1.5~2.5 ng/ml) during the surgery
  Interventions: Drug: remifentanil infusion group

INTERVENTIONS:
Drug: dexmedetomidine infusion group — dexmedetomidine as anaesthetic adjuvant
  Arms: dexmedetomidine infusion group
Drug: remifentanil infusion group — remifentanil as anaesthetic adjuvant
  Arms: remifentanil infusion group

SUMMARY:
This study was performed to compare the effect on of a postoperative sore throat between dexmedetomidine and remifentanil in patients undergoing thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled primary thyroidectomy were enrolled and their physical status was American Society of Anesthesiologists (ASA) class 1 or 2

Exclusion Criteria:

* Patients with respiratory tract disease, previous head, and neck surgery, preexisting steroid or non-steroidal anti-inflammatory drug use, and known or suspected difficult airway

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative sore throat at rest | 6 hours after surgery
  0=none; 1=occur
incidence of postoperative sore throat at swallowing | 6 hours after surgery
  0=none; 1=occur
severity of postoperative sore throat at rest | 6 hours after surgery
  4-point scale (0=none; 1=mild; 2=moderate; 3=severe)
severity of postoperative sore throat at swallowing | 6 hours after surgery
  4-point scale (0=none; 1=mild; 2=moderate; 3=severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Eun kyung Choi, Daegu, Korea (the Republic Of), South Korea

IPD SHARING:
Plan to Share IPD: Yes